CLINICAL TRIAL: NCT00654472
Title: Quantification of Rheumatic Mitral Stenosis With Cardiac Magnetic Resonance Imaging and Comparison With Transthoracic Echocardiography
Brief Title: Mitral Valve Area Assessment: Comparison With Transthoracic Echocardiography and Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Florence Nightingale Hospital, Istanbul (Other)
Responsible Party: Prof. Dr. Saide Aytekin, T.C. Istanbul Bilim University, Florence Nightingale Hospital
Other Study IDs: OY1975
Record Dates: First submitted 2008-04-02; First posted 2008-04-08 (Estimated); Last update posted 2008-04-08 (Estimated); Status verified 2008-04

CONDITIONS: Mitral Valve Stenosis
Keywords: magnetic resonance imaging, mitral valve area
MeSH Terms: conditions — Mitral Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Mitral valve area above 1.5 cm2
- B: Mitral valve area 1.5 cm2 and below 1.5 cm2

SUMMARY:
To compare mitral valve area in rheumatic mitral valve stenosis with cardiac magnetic resonance imaging and conventional transthoracic echocardiography.

DETAILED DESCRIPTION:
Clinical assessment of severity of mitral stenosis depends on both the presence of symptoms and mitral valve area . Evaluation of mitral valve area with transthoracic echocardiography maintains rapid, accurate analysis of valve disease and serves as a practical gold standard for clinical evaluation. Cardiac magnetic resonance imaging (CMRI) is a recently used method that allows to evaluate cardiac structures and function noninvasively. Direct visualization of valve area with CMRI is also possible and it has been shown that the valve area assessed by CMRI planimetry correlates reliably with the invasive assessment. Velocity-encoded cardiac magnetic resonance imaging can be used to quantify mitral valve area. The objective of this study was to evaluate mitral valve area with CMRI and compare it with echocardiographic methods including 2D planimetry, Doppler continuation equation and Doppler pressure half-time

ELIGIBILITY:
Inclusion Criteria:

* rheumatic mitral valve stenosis

Exclusion Criteria:

* Degenerative mitral valve disease
* EF<50%
* atrial fibrillation
* inconclusive planimetric assessment
* moderate or severe mitral regurgitation
* moderate or severe aortic regurgitation
* history of previous mitral valve commissurotomy or balloon valvotomy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-06 (Estimated); Study Completion 2008-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Saide Aytekin, Professor, Study Director — T.C. Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology
Locations (2):
- Turkey (Türkiye) (2):
  - Florence Nightinngale Hospital, Istanbul
  - TC.Istanbul Bilim University, Florence Nightingale Hospital, Division of Cardiology, Istanbul

REFERENCES:
- [Background] Lin SJ, Brown PA, Watkins MP, Williams TA, Lehr KA, Liu W, Lanza GM, Wickline SA, Caruthers SD. Quantification of stenotic mitral valve area with magnetic resonance imaging and comparison with Doppler ultrasound. J Am Coll Cardiol. 2004 Jul 7;44(1):133-7. doi: 10.1016/j.jacc.2004.03.038. PMID 15234421
- [Background] Djavidani B, Debl K, Lenhart M, Seitz J, Paetzel C, Schmid FX, Nitz WR, Feuerbach S, Riegger G, Luchner A. Planimetry of mitral valve stenosis by magnetic resonance imaging. J Am Coll Cardiol. 2005 Jun 21;45(12):2048-53. doi: 10.1016/j.jacc.2005.03.036. PMID 15963408